CLINICAL TRIAL: NCT00384709
Title: Geriatric Education and Its Effect on Certain Aspects of Hospital Care of the Nursing Home Patients
Brief Title: Geriatric Education and Its Effect on Certain Aspects of Hospital Care of Nursing Home Patients
Status: Completed | Type: Observational
Sponsor: Maimonides Medical Center (Other)
Responsible Party: Sergey I Genkin, MD, Maimonides Medical Center
Other Study IDs: gerivsnot
Record Dates: First submitted 2006-10-03; First posted 2006-10-06 (Estimated); Last update posted 2011-08-18 (Estimated); Status verified 2011-08

CONDITIONS: Frail Elderly; Patient Care
Keywords: Elderly; Hospitalization; Geriatrics; Mortality; Readmission; Length of Stay

SUMMARY:
Nursing home patients admitted to the hospital pose a significant challenge for health care providers. Geriatric teaching pays particular attention to these admissions and related problems. However, it is yet to be proven, whether geriatric training helps to overcome any of these issues in a better way than through non-geriatric education. The study aims to prove that geriatric training provides advantages over non-geriatric training in caring for nursing home patients admitted to the hospital.

DETAILED DESCRIPTION:
Context: Nursing home patients admitted to the hospital pose a significant challenge for health care providers. Geriatric age, frailty, multiple readmissions, prolonged length of stay, and high mortality are just a few attributes of nursing home patients in the hospital. Geriatric teaching pays particular attention to these challenging problems. However, it is yet to be proven, whether geriatric training helps to overcome any of these issues in a better way than through non-geriatric education.

Objective: To test the hypothesis that geriatric care provides advantages over non-geriatric training in caring for nursing home patients admitted to the hospital in regards to length of stay, rate of expirations and rate of readmissions. The secondary objective is to compare expirations and readmissions among patients cared for by geriatricians and non-geriatricians.

Design, Setting, and Participants: Retrospective cohort study of patients admitted from Metropolitan Jewish Geriatric Nursing Home (MJGNH) to Maimonides Medical Center (MMC) over a certain period of time and under the care of geriatricians, non-geriatric internists, and surgeons. Comparison of the three study groups by age, sex, expiration rate, length of hospital stay (LOS) and readmission rate. Comparison of expired patients by age, sex and average LOS. Comparison of readmissions, expiration rate, by preservation of continuity of care, and by emergency room visits without admission.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to Maimonides Medical Center (MMC) from affiliated Metropolitan Jewish Geriatric Nursing Home (MJGNH) for a 3 month period.

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: - All patients admitted to Maimonides Medical Center (MMC) from affiliated Metropolitan Jewish Geriatric Nursing Home (MJGNH) for a 3 month period.
Sampling Method: Non-Probability Sample
Dates: Start 2006-09; Study Completion 2007-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sergey I Genkin, MD, Principal Investigator — Maimonides Medical Center